CLINICAL TRIAL: NCT06484322
Title: Strategies Empowering Activities in Everyday Life (SEE 2.0); A Feasibility Evaluation of an Internet-based Occupational Therapy Intervention
Brief Title: Strategies Empowering Activities in Everyday Life: An Internet-based Occupational Therapy Intervention
Acronym: SEE2:0
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luleå Tekniska Universitet (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEE-633 940
Record Dates: First submitted 2024-06-20; First posted 2024-07-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-01

CONDITIONS: Chronic Disease
Keywords: Chronic disease; Self-management; Activities of daily life; Internet-based; Tele-rehabilitation; E-health; Occupational therapy; Prevention; Rehabilitation; Long-term health conditions
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The feasibility study has been designed as a longitudinal pre-test, post test trial without a control group embedded in a mixed method approach. The participants will receive the internet-based occupational therapy intervention 'SEE'.
  Data from the participants will be collected at baseline (0) and 4- and 12 months post baseline.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The group will receive the internet-based intervention 'SEE' focusing on supporting self-management of activities in everyday life to promote health. Beside SEE, they will also receive care as usual.
  Interventions: Behavioral: Strategies Empowering Activities in Everyday life (SEE 2.0)

INTERVENTIONS:
Behavioral: Strategies Empowering Activities in Everyday life (SEE 2.0) — SEEs internet-based intervention process begins with supporting the client to explore the need of and readiness for changes in everyday life. Thereafter, the client is supported to self-analyse their engagement in activities in everyday life along with use of management strategies in everyday life. Next, the client takes on web- modules including short educational movies with subsequent analyses and reflections. The modules aim to support the development of self-management by improving the knowledge of how strategies and changes in daily activities can prevent disabilities and contribute to improved health. After that, the focus is on establishing an activity plan with goals and activity-based management strategies to promote an active everyday life. The clients' implementation of the plan is supported through follow-up meetings. During the whole intervention process, the client is regularly supported by an occupational therapist through feedback and online guiding dialogues.

SUMMARY:
The purpose of the study is to evaluate the feasibility, potential outcomes and the implementation process of a second updated version of an internet-based intervention in occupational therapy, focusing on self-management in activities of everyday life to promote health in people with chronic diseases.

DETAILED DESCRIPTION:
The number of people with chronic disease is increasing as is the need of preventive efforts to facilitate their health. Chronic diseases are defined as 'long-term health conditions' that require constant attention and/or limit activities of daily living. People living with one or multiple chronic diseases experience difficulties to live an active everyday life and restrictions of engagement in various activities are common. Interventions that support their process of change and development of self-management in everyday life in relation to their changed capacity needs to be established. Research shows that the access to interventions is facilitated by the use of internet-based solutions. Hence, an internet-based occupational therapy intervention 'Strategies Empowering activities in Everyday life' (SEE) has been developed that will be evaluated in a feasibility trial.

The feasibility study is designed as a longitudinal trial with pre-test, post test evaluation without control group embedded in a mixed method approach. Data will be collected by assessment tools, qualitative interviews and group interviews. Evaluation of the feasibility of the intervention and the study design will be conducted in terms of acceptability, adherence, values, and implementation, from the perspective of patients with chronic disease and health care personnel at different organizational levels in primary care, as well as in out-patient and in-patient care at a regional hospital.

The results from this feasibility study will support the continued development of SEE in future larger-scale evaluation studies. The goal is that SEE will add to existing interventions and becomes implemented in clinical practice. The results will be published in peer-reviewed scientific journals and presented at conferences.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with, or at risk of developing, a chronic disease/long-term condition such as long-term pain, stress-related conditions, chronic fatigue syndrome, rheumatological diseases, lung diseases, or neurological conditions.
* Age: 18-75 years
* Experiencing difficulties to have an active everyday life and/or experiencing a need to develop self-management strategies in everyday life.
* Have access to a screen/computer, internet and e-ID as well as being able to use them
* Be able to participate in the program, including be ready for a process of change
* Understanding of the Swedish language in written and oral form.

Exclusion Criteria:

* Sickness or disease which causes difficulties with understanding written and verbal advice (e.g. mental or cognitive illness).
* Having an ongoing misuse
* Receiving palliative care

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The Satisfaction with Daily Occupation (SDO-13) | Change from baseline to four- and twelve months post-base line
  Measures change in satisfaction of daily occupations through a structured interview with 13 questions within areas such as work/studies, leisure, home and self-care occupations. Satisfaction with occupations is measured on an ordinal scale with a score ranging from 0-7. The total rating range between 13-91. Higher score indicates a higher satisfaction with daily occupations.
Occupational Balance Questionnaire (OBQ) | Change from baseline to four- and twelve months post-base line
  Measures change in perceived occupational balance; occupational balance reflects a person's subjective perception of having the right amount of- and the right variation between activities. The OBQ consist of 11 items rated on a four-point ordinal scale, scored 0 to 3. A total score may range between 0 and 33 where a higher score implies a higher sense of occupational balance.
Occupational values with pre-defined items (Oval-pd). | Change from baseline to four- and twelve months post-base line
  Measures change in occupational values which reflects the subjective perception of concrete, symbolic or self-rewarding values in activities. The Oval-pd consists of 18 items rated on a four-point ordinal scale, scored 1 to 4. The responses add up to a total score between 18-72, a higher score indicates higher occupational value in the activities of everyday life.

SECONDARY OUTCOMES:
Life satisfaction questionnaire (Lisat-11) | Change from baseline to four- and twelve months post-base line
  Measures a change in life satisfaction. Lisat-11 consists of 11 items rated on an ordinal scale scored 1-6. A higher score indicates a higher level of life satisfaction.
Work ability index (WAI) | Change from baseline to four- and twelve months post-base line
  Measures a change in self-perceived work ability. Self-perceived work ability is rated on a 10-point ordinal scale and a higher score indicates higher perceived work ability.
RAND-36 | Change from baseline to four- and twelve months post-base line
  Measures change in perceived health and function in everyday life and consists of 36 items with an ordinal scale across 8 dimensions of health. The dimensions of health are graded on a scale 0-100 and a higher score indicates a higher perceived health and function in everyday life.
General Self-Efficacy (GSE-10) | Change from baseline to four- and twelve months post-base line
  Measures change in self-reported self-efficacy which consists of 10 items on an ordinal scale from 1-4. The total score ranges from 10-40 and a higher score indicates higher self- efficacy.
Mental Fatigue Scale (MFS) | Change from baseline to four- and twelve months post-base line
  Measures change in perceived mental fatigue and consists of 14 items rated on an ordinal scale (0-3). The summarized score ranges from 0-42. Scores over 10.5 indicate fatigue.
EuroQol 5 Dimensions (EQ-5D) Thermometer | Change from baseline to four- and twelve months post-base line
  Measures a change in perceived health with a score ranging from 0-100. A higher score indicates better perceived health.
Perceived Stress Scale (PSS) | Change from baseline to four- and twelve months post-base line
  Change in perceived stress on 10 items rated on an ordinal scale (0-4). The summarised score range from 0-40. A higher score indicates a higher level of perceived stress.

OTHER OUTCOMES:
The experience of people with chronic conditions participating in the intervention process of SEE. | Repeated interviews during the intervention process, one- and four months post-baseline
  Qualitative individual open-ended interviews with client participants focusing on experiences of SEEs intervention process.
The acceptability and value of SEE from the perspective of the clients. | Four months post-baseline
  A study specific questionnaire. The items are rated on an ordinal scale, ranging from 1 to 4. Higher scores reflect higher levels of acceptability and value of SEE.
The adherence to SEE. | Through intervention completion, an average of 1 year
  The adherence of SEE will be studied with a structured interview using a study specific feasibility registration form assessing whether the intervention is delivered and taken as intended. The structured individual interview based on the feasibility registration form will be conducted with the occupational therapist delivering SEE to each client.
The experience of how feasibility, implementation, and context influence SEE. | Through study completion, an average of 2 year
  Experiences the feasibility and the implementation process of SEE from the perspectives of the delivers, i.e., the occupational therapists, their managers and other stakeholders/key persons will be explored qualitatively in groups interviews.
Number of participants recruited retention and drop-out rates. | Through study completion, an average of 2 year
  The recruitment process and resulting sample will be studied by the use of study-specific registration forms.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Larsson Lund, Professor, Study Chair — LTU
Locations (2):
- Sweden (2):
  - Luleå university of technology, Luleå, None Selected
  - Luleå University of Technology, Luleå

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsson-Lund M, Karlsson Sundbaum J, Mansson Lexell E, Spinord L. Feasibility study of the internet-based intervention 'Strategies for Empowering activities in Everyday life' (SEE 2.0) for use by people with chronic diseases and long-term disorders in healthcare: a study protocol. BMJ Open. 2025 Oct 21;15(10):e102026. doi: 10.1136/bmjopen-2025-102026. PMID 41125291